CLINICAL TRIAL: NCT06310694
Title: Does Fixing Peripheral Intravenous Catheter With Additional Circular Dressing Material Reduce PIVC Failure And Complications? A Randomized Controlled Trial
Brief Title: Additional Circular Dressing Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Şeyma Turan, PhD, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGE-HEM-SL-01
Record Dates: First submitted 2024-02-16; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Nurse's Role
Keywords: peripheral cannulation; catheter related complications; infusions; intravenous; dressing; nursing

STUDY DESIGN:
Intervention Model Description: In our study, a comparison was made of PIVCs applied to patients in the control (fixation of PIVC with a sterile transparent dressing) and intervention (fixation of PIVC with a sterile transparent dressing and application of an elastane circular dressing on it) groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Elastane circular dressing on sterile transparent dressing) (Experimental): A peripheral intravenous catheter was placed by following all the steps applied to the control group. A circular dressing made of elastane material was placed on the patients in the intervention group on a sterile transparent dressing to provide additional fixation on the peripheral intravenous catheter. There is no need to remove additional circular dressings during intravenous therapy.
  The peripheral intravenous catheter was monitored for 72 hours with 8-hour observations. Peripheral intravenous catheter was evaluated for infiltration, phlebitis, pain, obstruction, dressing stability, and leakage.
  Interventions: Combination Product: intervention group (Elastane circular dressing on sterile transparent dressing)
- Control group (fixation of PIVC with a sterile transparent dressing) (No Intervention): Peripheral intravenous catheter application was performed by the researcher in accordance with all steps. In the study, only patients who received a 20-gauge peripheral intravenous catheter were followed. The patient's peripheral intravenous catheter was fixed by the researcher with a sterile transparent dressing.
  The peripheral intravenous catheter was monitored for 72 hours with 8-hour observations. Peripheral intravenous catheter was evaluated for infiltration, phlebitis, pain, obstruction, dressing stability, and leakage.

INTERVENTIONS:
Combination Product: intervention group (Elastane circular dressing on sterile transparent dressing) — A circular dressing made of elastane material was placed on the patients in the intervention group on a sterile transparent dressing to provide additional fixation on the peripheral intravenous catheter.
  Arms: Intervention Group (Elastane circular dressing on sterile transparent dressing)

SUMMARY:
The study was conducted to determine the effect of fixing peripheral intravenous catheter (PIVC) with additional circular dressing material on the duration of PIVC stay and complications related to peripheral intravenous catheterization. In our study, a comparison was made of PIVCs applied to patients in the control (fixation of PIVC with a sterile transparent dressing) and intervention (fixation of PIVC with a sterile transparent dressing and application of an elastane circular dressing on it) groups in a public hospital in Turkey. All-cause PIVC failure was significantly higher in the intervention group (70.2%) compared to the control group (45.5%). It has been determined that fixing the PIVC with additional circular dressing material prolongs the duration of PIVC stay at the site.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled study to determine the effect of fixing the peripheral intravenous catheter (PIVC) with additional circular dressing material on the duration of stay of the peripheral intravenous catheter and complications related to peripheral intravenous catheterization. In our study, a comparison was made of PIVCs applied to patients in the control (fixation of PIVC with a sterile transparent dressing) and intervention (fixation of PIVC with a sterile transparent dressing and application of an elastane circular dressing on it) groups in a public hospital in Turkey. In our study, PIVC failure was defined as PIVC removal before the end of treatment due to phlebitis, infiltration, accidental dislodgement, occlusion, and leakage. A total of 91 (47 intervention, 44 control) participants were included in the study between April 2023 and September 2023. All-cause PIVC failure was significantly higher in the intervention group (70.2%) compared to the control group (45.5%). It was determined that fixing the PIVC with additional circular dressing material prolongs the duration of PIVC stay at the site. It is recommended that this study be conducted with a different patient population and multicenter.

ELIGIBILITY:
Inclusion criteria

* Individuals between the ages of 18-65
* Literate individuals
* Individuals who can communicate and fully focus
* Individuals without vision, hearing or perception problems

Exclusion criteria

* Individuals hospitalized for less than 72 hours
* Individuals with edema degree 2 and above
* Individuals receiving Total Parenteral Nutrition, colloid, blood products
* Individuals with a BMI level of 29.9 and above (obese)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 91 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Skin Penetration Difficulty Rating Scale | four months
  The Numerical Rating Scale was used by the investigator who performed the peripheral intravenous catheterization attempt to evaluate the severity of difficulty penetrating the skin. It is a scale with numbers from 1 to 10, with 1 (easy) on one end and 10 (very difficult) on the other end. After PIVC application, the difficulty of penetrating the skin during catheter insertion was evaluated by the researcher, scoring between 1 and 10.
Visual Infusion Phlebitis Diagnostic Scale | four months
  Visual Infusion Phlebitis Diagnosis Scale includes grading steps and the symptoms of phlebitis seen at each stage in case of observation of the catheter for possible risks while applying treatment with a peripheral intravenous catheter or in case of phlebitis development. On this scale, symptoms of phlebitis such as redness, pain, swelling, fever and stiffness are rated from 1 to 5.
Infiltration Rating Scale | four months
  The infiltration rating scale is used to determine the development and extent of infiltration. On the infiltration scale, infiltration development is graded between 0 and 4 points.
Data Collection Form for the Patient Who Had a Peripheral Intravenous Catheter | four months
  In this form, information such as the patient's age, gender, weight, height, BMI (Body Mass Index), diagnosis, chronic disease, date and time of PIVC application, date and time of PIVC termination, reason for PIVC termination, and the region where PIVC was applied were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Khorshid, Prof. Dr., Study Director — Ege University
Locations (1):
- Şeyma Turan, Turgutlu, Manisa, Turkey (Türkiye)